CLINICAL TRIAL: NCT06949202
Title: The Effect of Diaphragmatic Breathing Exercises on Stress and Exam Anxiety in Final-Year High School Students During the Exam Period: "I Breathe, I Relieve"
Brief Title: Diaphragmatic Breathing Exercises on Stress and Exam Anxiety in High School Seniors: A Randomized Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igdir University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Sema Bugusan Oruc, Assistant Professor in the Department of Physiotherapy and Rehabilitation, Igdir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I1.25
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Test Anxiety; Diaphragmatic Breathing; Stress Measurement, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercises (Experimental): diaphragmatic breating breath control exercises
  Interventions: Other: breating exercises
- Control Group (No Intervention): Participants in this group will not receive any training during the intervention period. They will only undergo evaluations at baseline and 4 weeks later. To ensure ethical standards, respiratory training will be offered to this group after the study is completed.

INTERVENTIONS:
Other: breating exercises — diaphragmatic breathing
  Arms: Breathing Exercises

SUMMARY:
This study aims to evaluate the effect of diaphragmatic breathing exercises on stress and exam anxiety in final-year high school students during the exam period. The intervention, named "I Breathe, I Relieve," will include a series of controlled breathing exercises designed to reduce stress and anxiety symptoms. Participants will be asked to practice diaphragmatic breathing techniques daily for a specific period leading up to their exams. The study will measure changes in stress levels and anxiety through standardized scales and questionnaires, comparing results before and after the intervention. The study will contribute to understanding the impact of breathing exercises on mental health in young individuals facing academic pressures.

DETAILED DESCRIPTION:
This study will be conducted in the city of Iğdır, Türkiye, and will involve final-year high school students currently enrolled in educational institutions in the region. Necessary permissions will be obtained from the Iğdır Provincial Directorate of National Education prior to the study.

The project is supported by TÜBİTAK 2209-A - University Students Research Projects Support Program.

Parental meetings will be organized, during which detailed information about the study will be provided to the families. The study will begin six weeks prior to the national university entrance examination.

After obtaining informed consent from both students and their families, demographic data including age, height, weight, and socio-cultural background will be recorded.

Oxygen saturation levels will be measured using a pulse oximeter.

To assess exam anxiety levels, the Tex Anxiety Inventory (TAI) will be used. This scale, developed by Spielberger and adapted into Turkish, consists of 20 items and two subscales: Worry (8 items) and Emotionality (12 items). Each item is rated on a 4-point Likert scale ranging from "almost never" to "always". The inventory evaluates the level of anxiety and its components experienced by individuals (References 8, 9).

To measure perceived stress levels, the Perceived Stress Scale (PSS) will be administered. The PSS assesses the degree to which individuals perceive situations in their lives as stressful. It consists of 14 items scored on a 5-point Likert scale ranging from 0 (never) to 4 (very often), with total scores ranging from 0 to 56. Higher scores indicate higher perceived stress levels (Reference 10).

Following initial evaluations, participants will be randomly assigned to either an intervention group or a control group. The intervention group will receive training in diaphragmatic breathing, relaxation techniques, and respiratory exercises, including respiratory muscle training using a spirometer (References 4, 11).

These training sessions will be conducted once a week for 4 consecutive weeks, with each session lasting approximately 20 minutes. Oxygen saturation will be measured with a pulse oximeter before and after each session.

At the end of the 4-week intervention period, both the Test Anxiety Inventory and Perceived Stress Scale will be re-administered to assess changes in stress and anxiety levels. Statistical analyses will be conducted accordingly.

This is a randomized controlled trial (RCT). Students in the control group will undergo assessments but will not receive any training during the study period. However, to prevent ethical concerns, the same respiratory training will be offered to the control group participants after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant and their parent/legal guardian must provide informed consent.
* Must be a final-year high school student preparing for the national university entrance exam.
* Must be in good general health.No chronic illnesses that pose a risk for participation.
* Aged between 16 and 19 years.

Exclusion Criteria:

* Participant and/or their parent/legal guardian do not provide informed consent.
* Failure to fully complete data collection tools (questionnaires, forms, etc.).
* Inability to actively participate in the exercise sessions.
* Presence of chronic health conditions that contraindicate participation in respiratory exercises.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Exam Anxiety Level | Baseline and 4 weeks after intervention
  Change in scores on the Exam Anxiety Inventory from baseline to 4 weeks after intervention.
Change in Perceived Stress Level | Baseline and 4 weeks after intervention
  Change in scores on the Perceived Stress Scale (14-item version) from baseline to 4 weeks after intervention.

SECONDARY OUTCOMES:
Change in Oxygen Saturation | During each training session (weekly, over 4 weeks)
  Measured before and after each respiratory training session using pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: sema büğüşan oruç, Study Director — Iğdır Uni
Locations (1):
- Iğdır Uni, Iğdır, State, Turkey (Türkiye)

REFERENCES:
- [Result] Rosenberg A, Hamiel D. Reducing Test Anxiety and Related Symptoms Using a Biofeedback Respiratory Practice Device: A Randomized Control Trial. Appl Psychophysiol Biofeedback. 2021 Mar;46(1):69-82. doi: 10.1007/s10484-020-09494-9. Epub 2021 Jan 2. PMID 33389280